CLINICAL TRIAL: NCT05610696
Title: Effects of Different Modalities of Aquatic Physiotherapy on Biomechanical and Functional Behavior of Subjects With Knee Osteoarthrosis
Brief Title: Different Modalities of Aquatic Physiotherapy in Patients With Knee Osteoarthrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Fernanda Cechetti, Sponsor-Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FUHSPortoAlegreCesar
Record Dates: First submitted 2022-01-20; First posted 2022-11-09 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Hydrotherapy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial, of the crossover type
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low impact immersion (Experimental): This intervention will use the principles of Ai Chi, a model defined as a low-intensity aquatic exercise strategy
  Interventions: Other: Low impact immersion
- Conventional aquatic physiotherapy (Experimental): In this intervention, medium impact exercises will be performed, with a comfortable movement speed.
  Interventions: Other: Conventional aquatic physiotherapy
- High intensity aquatic physiotherapy (Experimental): In this intervention, high-impact exercises will be performed, with maximum movement speed, twice time of the medium-intensity protocol
  Interventions: Other: High intensity aquatic physiotherapy

INTERVENTIONS:
Other: Low impact immersion — Consists of a sequence of shoulder, trunk and hip movements. In this modality, the aim will be to understand the physiological effects of immersion in heat water. Resisted movements (either by turbulence or by floats) or interventional maneuvers in the knee joints will not be performed. Considering the period of 5 minutes for acclimatization to the liquid environment, the program will last approximately 47 minutes.
  Arms: Low impact immersion
Other: Conventional aquatic physiotherapy — include warm-up, strengthening and calming down activities. Aquatic steppes will be used to ensure that all participants will maintain the waterline level approximately in the xiphoid appendix. For strengthening activities, the exercises must be performed at an adequate speed, which ensures a comfortable level for the activity. For this purpose, a subjective feedback will be extracted from the participants constantly. The warm-up sequence consists of six different active hip and knee movements performed at maximum range of motion and contributes to neuromuscular activation. For strengthening, each movement should be performed for 1 minute (30 seconds for each lower limb) followed by a period of 30 seconds of rest between each movement.
  Arms: Conventional aquatic physiotherapy
Other: High intensity aquatic physiotherapy — In this modality subjects will perform the same sequence of exercises of the Conventional Aquatic Physiotherapy program will be respected. However the work load and speed will be adjusted to the maximum level. For strengthening, each movement should be performed for 2 minutes (1 minute for each lower limb) followed by a period of 30 seconds of rest between each movement. To guarantee the maximum effort of the participants, verbal stimuli will be constantly provided. The program will last approximately 68 minutes.
  Arms: High intensity aquatic physiotherapy

SUMMARY:
The aim of this study is to evaluate the effects of different modalities of aquatic physiotherapy on the biochemical and functional behavior of patients with knee's Osteoarthritis.

DETAILED DESCRIPTION:
The subjects will be informed about the study and its potentials risks and sign the informed consent. The sample will be submitted to three different modalities of AF interventions: (a) low impact immersion, (b) conventional aquatic physiotherapy and (c) high intensity aquatic physiotherapy. The functional variables of flexibility, pain, joint volume will be evaluated before and immediately after each intervention whereas the biochemical variables will be evaluated from the analysis of peripheral blood following times: baseline moment (immediately before the intervention), moment 1 (immediately after the intervention), and moment 2 (24 hours after the intervention).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 50 years old and diagnosed with OA in at least one knee
* Presence of pain and at least one functional dysfunction for at least 6 months
* Absence of physical limitation that prevents the exercise protocol from being performed
* Kellgren and Lawrence ranking between I and IV
* walk independently and without auxiliary device

Exclusion Criteria:

* Inflammatory, rheumatic or autoimmune conditions
* Use of psychotropic, immunosuppressive and steroid medications
* Antioxidant consumption
* Alcohol and tobacco consumption
* Progressive ankylosis states
* neurological injuries
* Infections or skin diseases that contraindicate swimming pool immersion
* Surgical procedures on the knee joint in the last 12 months (excluding meniscectomy or arthroscopy)
* Lower Limb Joint Prosthesis
* Presence of inflammatory or infectious diseases, uncontrolled systemic arterial hypertension, uncontrolled diabetes, chronic obstructive pulmonary disease and history of ischemic heart disease
* Self-report of aquatic phobia and chlorine allergies

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2023-12-03 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Biochemical variables over time | Baseline moment (immediately before the intervention), moment 1 (immediately after the intervention) measured in all interventions
  Variations in the concentration of and Glutathione perioxidase in peripheral blood resulting from three aquatic physical therapy interventions evaluated comparatively between the different interventions in U/L
Biochemical variables over time | Baseline moment (immediately before the intervention), moment 1 (immediately after the intervention) measured in all interventions in mg/mL
  Variations in the concentration of Metalloproetinase

SECONDARY OUTCOMES:
Degree of pain over time | Baseline moment (immediately before the intervention), moment 1 (immediately after the intervention) measured in all interventions.
  Performed using the visual analogue pain scale, from a scale graduated from zero to 10, in which zero corresponds to cases without pain and 10 corresponds to the worst imaginable pain.
Edema over time | Baseline moment (immediately before the intervention), moment 1 (immediately after the intervention)
  Performed based on the measurement of the circumference of the affected knee. Result expressed in centimeters
Flexibility over time | Baseline moment (immediately before the intervention), moment 1 (immediately after the intervention) measured in all interventions.
  Assessed by measuring the amplitude of the active and passive movement for the knee flexion and, for that, a conventional goniometer will be used. Result expressed in degrees
Muscle strength over time | Baseline moment (immediately before the intervention), moment 1 (immediately after the intervention) measured in all interventions.
  Measured by dynamometer to assess knee extension strength. Results expressed in kg of force.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Augusto Teixeira C, Haas L, Frata B, Fiori Bortoli A, Scalco Acco F, de Castro G, Cechetti F. Effects of a low, medium, and high-intensity aquatic physiotherapy protocol on functional and biochemical parameters in individuals with knee osteoarthritis: protocol for a crossover randomized controlled trial. F1000Res. 2024 Sep 16;12:1605. doi: 10.12688/f1000research.140342.4. eCollection 2023. PMID 39296351